CLINICAL TRIAL: NCT07153939
Title: Multicenter Pivotal Study of the Velocity™ Percutaneous Arterio-Venous Fistula System
Brief Title: Pivotal Study of the Velocity™ pAVF System
Acronym: VENOS-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venova Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0865
Record Dates: First submitted 2025-08-20; First posted 2025-09-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Hemodialysis Access; Arteriovenous Fistula; End Stage Renal Disease (ESRD)
Keywords: percutaneous AVF; pAVF; endovascular AVF; endoAVF; Arteriovenous Fistula; AVF; VENOS-3; VENOS3
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Velocity pAVF System Treatment Arm (Experimental): Participants in this single-arm, open-label study will undergo creation of a dialysis access using the Velocity Percutaneous Arteriovenous Fistula (pAVF). The Velocity pAVF is designed to create an arteriovenous fistula (AVF) using a minimally invasive, catheter-based procedure through the skin, rather than open surgery. All subjects enrolled will receive the Velocity pAVF procedure. After the procedure, participants will be followed with physical examinations, duplex ultrasound, and dialysis assessments to evaluate fistula maturation, usability for hemodialysis, and long-term function. Additional procedures, if needed to assist maturation or maintain access function, will be recorded. Safety will be monitored throughout the study, including assessment of device-related and procedure-related complications.
  Interventions: Device: Velocity Percutaneous Arteriovenous Fistula

INTERVENTIONS:
Device: Velocity Percutaneous Arteriovenous Fistula — The Velocity pAVF is a catheter-based device used to create an arteriovenous fistula for hemodialysis access through a minimally invasive, percutaneous procedure. Unlike surgical AVF creation or other pAVF systems, Velocity is designed to simplify the procedure and improve consistency of maturation and long-term function. All participants in this study will undergo AVF creation using the Velocity pAVF.
  Other Names: Velocity pAVF

SUMMARY:
This study will evaluate the Velocity Percutaneous Arteriovenous Fistula (pAVF) System, a new minimally invasive method for creating dialysis access. People with kidney failure often require dialysis, which depends on having a reliable arteriovenous fistula (AVF). Traditionally, AVFs are created with surgery, but surgery can involve incisions, longer recovery, and sometimes additional procedures before the AVF can be used.

The Velocity System is designed to create an AVF through a small puncture in the skin using a catheter-based approach, without open surgery. This pivotal study will assess how safe the procedure is and how well it works for patients who need dialysis.

The study will take place at multiple centers in the United States and will enroll adults with kidney failure who are candidates for fistula creation. Participants will undergo the Velocity procedure and then be followed closely with exams, ultrasounds, and dialysis assessments for up to five years.

Taking part is voluntary. Patients may benefit from a less invasive approach to dialysis access, but the main goal is to collect information that could improve future care for people with kidney failure.

ELIGIBILITY:
Inclusion Criteria:

1. ESRD requiring hemodialysis access or CKD with anticipated need for hemodialysis within 6 months
2. Cubital perforating vein diameter ⩾ 2.0 and ⩽ 5.0 mm
3. Proximal radial artery diameter ⩾ 2.0 and ⩽ 4.0 mm
4. Age > 18 years and < 80 years
5. Willing and competent to give written informed consent
6. Willing and able to complete all study assessments and follow-up requirements

Exclusion Criteria:

1. Study extremity systolic blood pressure < 100mmHg
2. Subjects with occlusion of the ulnar or radial artery at any level or an abnormal Allen's test
3. Subjects with a previous ipsilateral arterio-venous graft or previous ipsilateral upper arm AVF.
4. Distance between Cubital Perforating Vein and Proximal Radial Artery > 3.0 mm
5. Cephalic vein diameter < 2.5 mm at any point from the CPV to the axillary vein
6. Central venous occlusion ipsilateral of the study extremity
7. Severe calcification of the radial artery that significantly impairs ultrasound visualization (e.g., acoustic shadowing) and thus precludes safe or accurate device deployment.
8. Evidence of active systemic infections or localized to the procedure access site within the past 7 days
9. History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months prior to study entry, ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
10. Any contraindication to antiplatelet therapy
11. Currently being treated with another investigational device or drug
12. Known adverse effects to sedation and/or anesthesia which cannot be adequately pre-medicated
13. Uncontrolled or poorly controlled diabetes defined as a HbA1C > 10%
14. Known hypercoagulable condition, bleeding diathesis or coagulation disorder
15. Lymphedema of the study extremity
16. Scheduled kidney transplant within 6 months of enrollment
17. Peripheral white blood cell count < 1,500 cells/μL or > 13,000 cells/μL and neutrophil > 80%
18. Platelet count < 75,000 cells/ μL
19. Current diagnosis of carcinoma (unless in remission > 1 year)
20. Pregnant or currently breast feeding
21. Allergies to nickel or nickel titanium alloy (NiTi) or any of the components of the Velocity Implant or Delivery System
22. Any other medical condition that in the opinion of the investigator would put the welfare of the subject at risk or confound interpretation of the study data
23. Investigator determines that vascular anatomy at intended index procedure site is inappropriate for use of investigational device prior to attempting needle access.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Physiologic Maturation | 6 weeks
  The proportion of participants that reach the binary outcome of Physiologic Maturation. Physiologic Maturation is a composite measure, reached when Duplex ultrasound demonstrates a brachial artery blood flow of ≥ 500 ml/min and an outflow vein diameter of ≥ 5 mm.
Serious Adverse Device Effect | 30 days
  Any Serious Adverse Event that reasonably suggests is caused by the device or procedure

SECONDARY OUTCOMES:
Functional Maturation | 6 months
  The number of participants with successful two needle cannulation for 75% of dialysis sessions over a consecutive 4 weeks period following pAVF creation
Unassisted Functional Maturation | 6 months
  The number of participants that reach functional maturation without any endovascular or surgical interventions to facilitate maturation and/or manage complications
Physiologic Maturation | 3 months
  The proportion of participants that reach the binary outcome of Physiologic Maturation. Physiologic Maturation is a composite measure, reached when Duplex ultrasound demonstrates a brachial artery blood flow of ≥ 500 ml/min and an outflow vein diameter of ≥ 5 mm.
Time to First Hemodialysis | Through 12 month follow up, on average at 3 months
  The interval from the time of pAVF creation to the first hemodialysis session using 2-needles in the ESRD subgroup
Number of Catheter Days | Through 12 month follow up, on average at 3 months
  The number of days from pAVF creation to central venous catheter removal in the ESRD subgroup.
Access Circuit Primary Patency | Assessed up to 5 years
  The interval of time from access creation until the first occurrence of any reintervention to maintain or reestablish patency or until access thrombosis or abandonment.
Velocity pAVF Primary Patency | Assessed up to 5 years
  The interval of time from access creation until the first occurrence of reintervention or thrombosis directly attributable to a causative lesion within 5 mm of each end of the Velocity pAVF.
Access Circuit Cumulative Patency | Assessed up to 5 years
  The interval of time from access creation until the final abandonment of the access, inclusive of all successful interventions to maintain or restore patency
Technical Success | Immediately after the intervention
  The proportion of subjects with successful delivery of the implant between the perforating cubital vein and the radial artery, and removal of the delivery system, at the index procedure.
Procedural Success | Immediately after the intervention
  The proportion of subjects with intraprocedural duplex ultrasound demonstrating arterialized flow in the cephalic vein
Freedom from Reintervention | Assessed up to 5 years
  The duration from the time of access creation until the first occurrence of a reintervention required to maintain or restore patency of the pAVF
Total Reinterventions | Assessed up to 5 years
  The total number of reinterventions over the life of the access until abandonment or when the subject exits the study.
Freedom from Serious Adverse Events | Assessed up to 5 years
  Defined as the interval of time from access creation to the first occurrence of any serious adverse event.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Trinity Research Group, Dothan, Alabama
  - West Coast Kidney Institute Concord, Concord, California
  - Apex Research, Riverside, California
  - Vascular and Embolization Specialists, Cocoa, Florida
  - Azura Vascular Care Jacksonville, Jacksonville, Florida
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - Aqua Research, Houston, Texas
  - Humble Vascular Surgical Center, Humble, Texas
  - Fresenius Vascular Care San Antonio, San Antonio, Texas
  - San Antonio Surgical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Request for data will be accepted after study completion and final publication of results.